CLINICAL TRIAL: NCT06658769
Title: Use of Transcranial Magnetic Stimulation in the Prevention of Post-Operative Cognitive Dysfunction in Elderly with Mild Neurocognitive Disorder
Brief Title: Use of Transcranial Magnetic Stimulation in the Post-Operative Cognitive Dysfunction in Elderly
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Clarice Tanaka, Director of Physiotherapy Division, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 58398022.1.0000.0068; 6.796.500 (Registry Identifier: PARECER)
Record Dates: First submitted 2024-10-21; First posted 2024-10-26 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Postoperative Cognitive Dysfunction
Keywords: Transcranial Magnetic Stimulation; Postoperative Cognitive Dysfunction; Theta Burst Stimulation
MeSH Terms: conditions — Postoperative Cognitive Complications | interventions — Clinical Protocols

STUDY DESIGN:
Intervention Model Description: After patients are recruited according to the eligibility criteria during the medical screening at the first preoperative outpatient clinic visit or through active search on the waiting list, agree to participate in the protocol, fill out the safety questionnaire for the use of TMS and the transcranial electrostimulation application form, they will be randomized and allocated into two intervention groups different from the surgical group, based on a random table generated by the website www.randomization.com . The person responsible for the randomization stage will not have any other participation in the study. The group allocation will be confidential and the information regarding the patient group will be placed in opaque and numbered envelopes. Each envelope will be opened on the first day of the neuropsychological evaluation. Group 3, non-surgical control with cognitive impairment, will be automatically directed to active stimulation.
Who Masked: Participant, Outcomes Assessor
Masking Description: Double-Blind Randomized Clinical Trial, both participants and outcomes assessors will be blinded to active or sham stimulation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Pre-surgical intervention group (PREG) (Active Comparator): Participants in the Pre-surgical intervention group (PREG) will undergo active rTMS 15 days before surgery. The protocol will be intermittent theta-burst (iTBS), with 3 pulses applied at 50Hz and modulated at 5Hz for 2s, repeated every 10s for a total of 120s, totaling 300 pulses, with intensity at 80% of the MRL. The stimulated targets will be the left and right posterior parietal cortex (P3 and P4) and the left and right dorsolateral prefrontal cortex (F3 and F4), totaling 1200 pulses per day
  Interventions: Other: Theta Burst Stimulation
- Pre-surgical Control Group (PRECG) (Sham Comparator): Participants in the Pre-surgical Control Group (PRECG) will undergo simulated rTMS with a 90º coil tilt with the lower part facing the scalp 15 days before surgery. The protocol will be intermittent theta-burst (iTBS), with 3 pulses applied at 50Hz and modulated at 5Hz for 2s, repeated every 10s for a total of 120s, totaling 300 pulses, with intensity at 80% of the MRL. The stimulated targets will be the left and right posterior parietal cortex (P3 and P4) and left and right dorsolateral prefrontal cortex (F3 and F4), totaling 1200 pulses per day.
  Interventions: Other: Theta Burst Stimulation Sham
- Non-surgical Control Intervention Group (COG) (Active Comparator): Participants in the Non-Surgical Control Intervention Group (COG) will undergo active rTMS. The protocol will be intermittent theta-burst (iTBS), with 3 pulses applied at 50Hz and modulated at 5Hz for 2s, repeated every 10s for a total of 120s, totaling 300 pulses, with intensity at 80% of the MRL. The stimulated targets will be the left and right posterior parietal cortex (P3 and P4) and the left and right dorsolateral prefrontal cortex (F3 and F4), totaling 1200 pulses per day
  Interventions: Other: Theta Burst Stimulation

INTERVENTIONS:
Other: Theta Burst Stimulation — Transcranial Magnetic Stimulation (TMS): A non-invasive brain stimulation (NIBS) technique that involves modulating brain excitability and activity, which can increase or decrease depending on the parameters used. Theta Burst Stimulation (TBS) mimics the brain's natural firing patterns more closely and may have greater effects on cognitive performance.
  Other Names: Protocol
  Arms: Non-surgical Control Intervention Group (COG); Pre-surgical intervention group (PREG)
Other: Theta Burst Stimulation Sham — Theta Burst Stimulation simulated with 90º coil orientation with lower part external to the scalp.
  Other Names: Protocol
  Arms: Pre-surgical Control Group (PRECG)

SUMMARY:
Postoperative Cognitive Dysfunction (POCD) is a prevalent condition with significant clinical, social, and financial impacts on patients and healthcare services. The term POCD refers to any signs of new cognitive impairment that exceed the expected time for recovery from the acute effects of surgery and anesthesia. Mild Cognitive Impairment (MCI) is among the main risk factors and is defined as a small cognitive decline from the previous level of performance in one or more cognitive domains, without interfering with daily activities. Considering the aging population linked to an increase in the number of individuals with MCI and a growing demand for surgery, the identification of interventions that can prevent the occurrence of POCD is necessary. Non-invasive brain stimulation (NIBS) techniques such as TMS (Transcranial Magnetic Stimulation) are widely used in research and clinical practice and involve the modulation of excitability and brain activity, potentially improving the individual's cognitive performance. The aim of this study is to assess the efficacy of a Theta Burst rTMS protocol with few sessions in preventing postoperative cognitive dysfunction in elderly individuals with mild neurocognitive disorder. Methodology: This will be a randomized, blinded clinical trial with volunteers aged > 60 years, candidates for elective surgeries, who will be randomly allocated into 2 groups: the groups will receive real or sham TBS 15 days before surgery. There will be 3 intervention sessions, with a 72-hour interval between them. Outcome measures will be cognitive psychological assessment and Stroop Test cognitive task performance before and after transcranial magnetic stimulation, after surgery and at the 3-month follow-up. There will be a non-surgical control group with cognitive impairment according to the study inclusion criteria and will receive active stimulation.

DETAILED DESCRIPTION:
Postoperative Cognitive Dysfunction (POCD) is a highly prevalent condition with significant clinical, social, and financial impacts for patients and their communities. Postoperative (PO) cognitive impairments have generally been divided into short- and long-term disturbances. Delirium, a short-term disorder, is defined according to the Diagnostic and Statistical Manual of Mental Disorders V (DSM-V) as impairment in attention, awareness, and cognition, fluctuating throughout the day and affected by endogenous and exogenous factors. It has an incidence of 37-46%, differing depending on the type of surgical procedure performed, with reports of up to 51%. In contrast, the term POCD has been used to refer to any new signs of cognitive impairment that exceed the expected time for recovery from the acute effects of surgery and anesthesia, being considered long-term. Among hospitalized PO patients aged 60 years or older, rates of up to 40% have been observed. Considering the aging population linked to a growing demand for surgery, identifying factors that increase the risk of POCD is necessary, as age is the biggest risk factor. Mild Cognitive Impairment (MCI) is one of the main risk factors and is defined as cognitive decline from a previous level of performance in one or more cognitive domains (complex attention, executive function, learning and memory, language, perceptual-motor, or social cognition), based on the concern of the individual, caregiver, or clinician. However, these changes do not interfere with the ability to be independent in daily activities. The conversion rate from MCI to dementia is 10 to 15% per year, regardless of any possible influence from anesthesia and surgery. However, there is evidence that anesthesia and surgery may exacerbate the pathological mechanisms of Alzheimer's disease, which could potentially increase this conversion rate. Pre-existing brain, heart, or vascular diseases, low educational levels, and alcohol use are also frequent risk factors. Iatrogenic factors also seem to contribute to POCD. Some articles speculate that POCD in the elderly is attributable to the use of benzodiazepines (BZDs) and anticholinergics (ACs), while others suggest that POCD is independent of the type of surgery or anesthesia used and would result from pre-existing brain fragility. Although a transient fluctuation in cognition during the postoperative period is often not considered concerning, it is important to note that POCD predicts the onset of future dementia and may contribute to chronic neurodegeneration, particularly with repeated surgical procedures.PO cognitive changes can clearly lead to a loss of autonomy in the elderly, prolong hospital stays, generate high medical costs, and increase mortality, making it a serious health and social problem that cannot be ignored. Current theories on the underlying mechanisms of POCD highlight the role of inflammation and immune activation. Surgery itself induces inflammatory processes, localized and systemic expression of pro-inflammatory cytokines, and signaling molecules. Tissue damage after surgery triggers the release of IL-1 and TNF- from endothelial cells and phagocytes, whose elevated levels induce the production of IL-6, increasing the extent of tissue trauma and triggering a cascade of events. The formed inflammatory cascade and cytokine release reach the central nervous system and have a direct relationship with the hippocampus. This brain region contains the highest number of cytokine receptors, has the highest density of IL-1 receptors, and although physiological levels of this cytokine are essential for optimal memory and learning processes in the hippocampus, excessive levels have been associated with decreased cognitive function in animal models. The hippocampus seems especially vulnerable to the harmful effects of systemically elevated inflammatory mediators due to the high density of TNF- receptors and numerous other receptors on the surface of endothelial cells in this brain region. The mechanism underlying impaired learning and memory resulting from excessive levels of IL-1 and other inflammatory mediators in the hippocampus involves harmful effects on long-term potentiation (LTP) and neurogenesis in this brain region, as demonstrated in several animal models. The cognitive reserve is a protective factor for the development of PO cognitive changes and that its increased levels are strongly protective for the incidence of dementia; including higher levels of education, greater occupational complexity, premorbid IQ, and a preference for mentally stimulating leisure activities. Studies in cognitively healthy humans have also shown that physical exercise improved global cognition and was associated with increased gray matter volume, while cognitive exercise was associated with reduced memory loss. Non-invasive brain stimulation (NIBS) techniques are widely used in research and clinical practice, involving the modulation of brain excitability and activity, which can increase or decrease depending on the parameters used, such as transcranial magnetic stimulation (TMS). Numerous in vitro and in vivo experimental models provide evidence that repetitive TMS (rTMS) can enhance long-term potentiation (LTP). LTP is a lasting increase in signal transmission between two neurons resulting from synchronous stimulation. It is one of several phenomena contributing to synaptic plasticity. Memory is thought to be encoded by modifying synaptic strength, so LTP is widely considered one of the main cellular mechanisms underlying learning and memory. These improvements in neural plasticity are observed alongside enhanced performance on hippocampal-dependent cognitive measures. The fundamental basis for brain function is brain oscillations in various frequency ranges. Several studies provide evidence supporting the idea that modulating specific frequency oscillations can alter cognition in healthy individuals. Additionally, rTMS has been used to improve cognitive function through the same mechanism. Particularly, several studies suggest that focal rTMS may promote the alteration and synchronization of human brain oscillations and reveal changes in cognition. According to Hoy and colleagues, neural synchrony refers to the coordinated firing of connected brain regions, which is considered essential for the integration of neural networks and cognitive performance. In other words, rTMS may be an effective oscillatory alteration approach with the potential to improve specific cognitive functions such as attention and perception. New forms of rTMS have recently been developed, including Theta Burst Stimulation (TBS), a new accelerated form of stimulation that more closely mimics the brain's natural firing patterns and may have greater effects on cognitive performance. TBS sessions usually last only 3-10 minutes, compared to conventional rTMS sessions. Faster daily treatments with TBS can allow for increased treatment capacity and reduced costs per session. Improvements in cognitive function using intermittent Theta Burst (iTBS) compared to those using traditional rTMS have been found and may be due to endogenous oscillations. It is important to note that theta and gamma bands have been linked to working memory processes. Oscillations play a critical role in integrating the different brain regions necessary for working memory, with synchronous activity between prefrontal and posterior parietal regions associated with successful working memory encoding. Current findings are promising, revealing a more substantial effect of iTBS compared to the best conventional rTMS protocol investigated so far. These findings indicate that iTBS may be a more suitable and accelerated protocol for cognitive promotion in patients diagnosed with cognitive deficits related to diseases such as Alzheimer's disease and vascular cognitive impairment. However, further patient-based studies with cognitive deficits are needed to explore the effects of iTBS on cognition in real-world settings and different patients. Therefore, the goal of this project is to explore new approaches to postoperative cognitive dysfunction, focusing on its prevention using brain magnetic stimulation techniques. So far, no pre- and postoperative intervention studies have shown robust results in preventing this clinical condition.

ELIGIBILITY:
Inclusion Criteria:

1. Patients over 60 years old
2. Patients scheduled for elective surgeries of moderate or large scale and candidates for general or spinal anesthesia;
3. Patients who demonstrate possible or probable cognitive impairment based on pre-operative screening using the 10-CS (10-point cognitive screening) tool; - For Non-surgical Control Intervention Group, only the first and third criteria will be applied.

Exclusion Criteria:

1. Contraindications for the use of Transcranial Magnetic Stimulation (metal implants in the head, history of seizures or epilepsy, brain trauma or surgery, intracranial hypertension, and complications from exposure to magnetic fields);
2. Medical diagnosis of Major Neurocognitive Disorder (any form of dementia, regardless of the stage);
3. Indication for skull surgery;
4. Conditions that interfere with cognitive testing (presence of severe hearing and vision loss, inability to understand Portuguese);
5. Ongoing medication adjustments that affect cortical electrical activity (antidepressants, antipsychotics);
6. Difficulty attending treatment during the stipulated evaluation and follow-up period, whether due to socioeconomic or clinical reasons;
7. Anticipation of surgical scheduling;

Ages: 60 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in Verbal Learning | 1st evaluation: Baseline. 2nd evaluation: 2 days after the application of the active or sham iTBS protocol. 3rd evaluation: 15 days after surgery (surgical groups) or 20 days after the second evaluation (non-surgical group). 4th evaluation: 3 months afte
  Hopkins Verbal Learning Test (HVLT) - This test consists of a list of 12 words. After the examiner reads the list, the patient is asked to repeat as many words as possible in any order. This procedure is repeated two more times, and after 25 minutes, a delayed recall is requested. The score is based on the number of words recalled in the delayed recall.
Changes in Attention and Executive Function: | 1st evaluation: Baseline. 2nd evaluation: 2 days after the application of the active or sham iTBS protocol. 3rd evaluation: 15 days after surgery (surgical groups) or 20 days after the second evaluation (non-surgical group). 4th evaluation: 3 months afte
  Trail Making Test (A and B) - The test is divided into two parts: the first part (TMT A) involves simple visual search and motor speed, while the second part (TMT B) requires complex visual search due to the alternation of stimuli, thus assessing executive function performance. In part A, the person must connect numbered circles in ascending order. In part B, they must draw lines alternating between numbers in ascending order and letters in alphabetical order. The test evaluates not only selective and alternating attention but also complex visual tracking and motor dexterity (Part A) as well as executive processes (Part B). The time spent and the number of errors made in each part are assessed.
Changes in Attention and Processing Speed | 1st evaluation: Baseline. 2nd evaluation: 2 days after the application of the active or sham iTBS protocol. 3rd evaluation: 15 days after surgery (surgical groups) or 20 days after the second evaluation (non-surgical group). 4th evaluation: 3 months afte
  Stroop Test - The Stroop test assesses selective attention, the ability to maintain focus on a task, and the inhibition of the tendency to provide impulsive responses, as well as the speed of information processing. In this task, 99 trials are presented on a computer, featuring the words "green," "red," and "blue," displayed in their respective colors (or not). It measures the response time to name the colors of words that are colored in their actual color (congruent trials) or to state the colors of words with different colors (incongruent trials). It also evaluates the number of correct responses in the trials. Data will be synchronized using MATLAB software.
Changes in Motor Skills | 1st evaluation: Baseline. 2nd evaluation: 2 days after the application of the active or sham iTBS protocol. 3rd evaluation: 15 days after surgery (surgical groups) or 20 days after the second evaluation (non-surgical group). 4th evaluation: 3 months afte
  The Grooved Pegboard Test - This is a manual dexterity test consisting of a board with 25 holes of the same shape (similar to a keyhole) and size, but arranged in a random orientation, along with small pegs that must be placed into the holes following a predetermined order, using only one hand. The raw data corresponds to the time taken to complete the task, measured in seconds. The dominant hand is tested first, followed by the non-dominant hand.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Sao Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hoy KE, Bailey N, Michael M, Fitzgibbon B, Rogasch NC, Saeki T, Fitzgerald PB. Enhancement of Working Memory and Task-Related Oscillatory Activity Following Intermittent Theta Burst Stimulation in Healthy Controls. Cereb Cortex. 2016 Dec;26(12):4563-4573. doi: 10.1093/cercor/bhv193. Epub 2015 Sep 23. PMID 26400923
- [Background] Chou YH, Ton That V, Sundman M. A systematic review and meta-analysis of rTMS effects on cognitive enhancement in mild cognitive impairment and Alzheimer's disease. Neurobiol Aging. 2020 Feb;86:1-10. doi: 10.1016/j.neurobiolaging.2019.08.020. Epub 2019 Aug 27. PMID 31783330
- [Background] Begemann MJ, Brand BA, Curcic-Blake B, Aleman A, Sommer IE. Efficacy of non-invasive brain stimulation on cognitive functioning in brain disorders: a meta-analysis. Psychol Med. 2020 Nov;50(15):2465-2486. doi: 10.1017/S0033291720003670. Epub 2020 Oct 19. PMID 33070785
- [Background] Evered L, Scott DA, Silbert B, Maruff P. Postoperative cognitive dysfunction is independent of type of surgery and anesthetic. Anesth Analg. 2011 May;112(5):1179-85. doi: 10.1213/ANE.0b013e318215217e. Epub 2011 Apr 7. PMID 21474666
- [Background] Skvarc DR, Berk M, Byrne LK, Dean OM, Dodd S, Lewis M, Marriott A, Moore EM, Morris G, Page RS, Gray L. Post-Operative Cognitive Dysfunction: An exploration of the inflammatory hypothesis and novel therapies. Neurosci Biobehav Rev. 2018 Jan;84:116-133. doi: 10.1016/j.neubiorev.2017.11.011. Epub 2017 Nov 26. PMID 29180259